CLINICAL TRIAL: NCT05771090
Title: First Clinical Evaluation of a Novel Glucose Non-invasive Sensor Technology in Patients With Type 1 Diabetes: a Single-arm Pilot Study
Brief Title: First Clinical Evaluation of a Novel Glucose Non-invasive Sensor Technology in Patients With Type 1 Diabetes
Acronym: VAARA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DCB Research AG (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: VAARA study
Record Dates: First submitted 2023-02-28; First posted 2023-03-16 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus
Keywords: Volatile Organic Compounds; Hypoglycaemia
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Sokru device, prototype
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Participants in the study arm will undergo the study procedure which are different induced glycaemic states.
  Interventions: Device: Sokru device

INTERVENTIONS:
Device: Sokru device — Different induced glycaemic states in people living with diabetes (PwD).

SUMMARY:
The primary aim of this clinical study is to find signal characteristics of VOCs detected by Sokru device during fasting, insulin injection and after glucose intake and to find the association with blood glucose variation in variant states of glycemia and hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* T1D with MDI or CSII therapy >1 year
* Age 18 - 50 (inclusive)
* Caucasian ethnicity
* BMI between 18.5 and 24.9 kg/m2 (inclusive)
* Usage of a continuous glucose monitoring (CGM)

Exclusion Criteria:

* Pregnancy or breastfeeding
* History of cardiovascular diseases
* Diabetes-related comorbidities
* HbA1c >9 %
* Epilepsy
* Known sensitivity to medical grade adhesives or other skin-related complications, which might influence the outcome
* Known sensitivity to Latex
* Participation in another investigation with an investigational drug within the 30 days preceding and during the present investigation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Characteristics of volatile organic compound (VOC) signals measured by the Sokru device | During the study procedure (approximately 5 hours)
  The primary outcome are changes in VOC signals measured by the Sokru at low glucose levels (below 3.0 -3.9 mmol/L) or during the time when the blood glucose level is decreasing (from 10 and 3.9 mmol/L).

SECONDARY OUTCOMES:
Volatile Organic Compound Signals | During the study procedure (approximately 5 hours)
  VOC signals measured by the Sokru device at different blood glucose levels
Blood glucose concentration | During the study procedure (approximately 5 hours)
  Blood glucose levels are measured with the continuous glucose measurement system and in the venous blood at the time of the appearance of VOC signal peaks or drops
Time of onset of subjective symptoms of hypoglycemia | During the study procedure (approximately 5 hours)
  Self-reported onset of subjective symptoms of hypoglycemia
Heart rate | During the study procedure (approximately 5 hours)
  Heart rate is measured with a Mindray device
Oxygen saturation | During the study procedure (approximately 5 hours)
  Oxygen saturation is measured with a Mindray device

CONTACTS AND LOCATIONS:
Overall Officials: Derek Brandt, Study Chair — DCB Research AG
Locations (1):
- Universitätsklinik für Diabetologie, Endokrinologie, Ernährungsmedizin & Metabolismus (UDEM) Inselspital, Universitätsspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No